CLINICAL TRIAL: NCT01927692
Title: Exploratory Study Of Immunological Profiles In Myasthenia Gravis Subjects That Receive Therapeutic Plasma Exchange
Brief Title: Therapeutic Plasma Exchange in MG
Acronym: TPE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00043906
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Myasthenia Gravis
Keywords: MG
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MG subjects: MG subjects will have serum acetylcholine receptor (AChR) antibodies
  Interventions: Other: Skin biopsy; Other: Single Fiber Electromyography

INTERVENTIONS:
Other: Skin biopsy — An optional skin biopsy will be performed in up to 5 subjects at baseline and 2 weeks after therapeutic plasma exchange is completed.
Other: Single Fiber Electromyography — An optional SFEMG study will be performed at baseline and 2 weeks after therapeutic plasma exchange is completed.
  Other Names: SFEMG

SUMMARY:
The primary objective of the study is to longitudinally profile immunoglobulin levels and autoantibody levels in subjects with myasthenia gravis (MG) who receive therapeutic plasma exchange (TPE).

DETAILED DESCRIPTION:
This is a prospective, multi-center, pilot biomarker study in subjects receiving TPE for the treatment of MG. No study medications will be given.

Ten (10) AChR antibody positive MG subjects will be enrolled in the study at 2 sites. Of these 10 MG subjects, up to 5 may be receiving chronic TPE.

The study period will be approximately 3 months and will consist of:

* Screening/baseline visit,
* TPE visit where subjects will undergo clinical evaluations and blood draws for immunological assays,
* End of TPE visit where information on the TPE procedure will be recorded, clinical measurements will be performed, and a blood sample will be drawn.
* Post-TPE period where subjects will undergo clinical evaluations and blood draws for immunological assays at week 1, week 2, week 3, week 6, and week 12 after TPE.

Study procedures performed outside of usual care will include optional single-fiber electromyography (SFEMG) studies, blood draws and optional skin biopsies.

ELIGIBILITY:
Inclusion Criteria:

* has the capacity to understand and sign an informed consent form
* 18 years or older
* diagnosis of MG based on clinical features
* has detectable serum autoantibodies to AChR
* has a clinical indication for the use of TPE to treat MG

Exclusion Criteria:

* unable or unwilling to comply with study procedures that include multiple venipunctures
* weighs less than 50Kg
* has a contraindication to treatment with TPE (e.g. clinically significant bleeding disorder)
* has muscle specific tyrosine kinase or low-density lipoprotein receptor-related protein 4 (LRP4) antibody positive MG
* has prior or current history of thymoma
* had a thymectomy in the past 6 months
* has received rituximab in the past 12 months
* has another coexisting autoimmune disease that is not clinically controlled or may preclude accurate study assessments according to the judgment of the PI
* has current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, or central nervous system disease
* has participated in an interventional clinical trial with a novel therapeutic agent in the past 6 months
* is cognitively impaired, a prisoner, or otherwise institutionalized at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially eligible subjects with MG that will receive TPE as part of their clinical care will be identified from clinic encounters, emergency department visits, and hospitalizations.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Immunoglobulin levels | 14 weeks
  Immunoglobulin and IgG subtype levels, AChR autoantibody levels, IgG/autoantibody ratio will be listed, summarized and plotted graphically by visit.

SECONDARY OUTCOMES:
Lymphocyte subpopulations | 14 weeks
  Peripheral blood mononuclear cells (PBMC) will be analyzed using highly standardized polychromatic flow cytometric techniques for the expression of a broad array of phenotypic markers. A B-cell and T-cell panel will be used to profile specific marker expression among PBMCs and define lymphocyte subpopulations.
SFEMG | 14 weeks
  The extensor digitorum communis muscle will be studied in every subject and the muscle tested must have increased jitter at the initial study. If examination of the extensor digitorum communis is not feasible or the jitter is normal at the initial study, the muscle to study will be at the discretion of the investigator performing the SFEMG test, preferably frontalis. In each SFEMG study, jitter from 20 paired muscle fiber potentials will be recorded whenever feasible. Recorded variables will include total number of muscle fiber pairs studied, abnormal muscle fiber pairs, blocking pairs, and mean consecutive difference (MCD).
Vaccination/protective antibodies | 14 weeks
  The time course for recovery of selected protective antibody levels removed during TPE will be summarized.
Clinical Outcomes Assessments | 14 weeks
  All clinical outcomes assessments data (MG-Composite, MG-ADL, MG-QOL-15, MG-MMT) will be listed and summarized by visit. Scores may be presented graphically. Immunological measurements will be correlated with clinical scores, if appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Guptill, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina